CLINICAL TRIAL: NCT00873327
Title: Pharmacokinetics and Safety of Piperacillin-tazobactam in Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Assistant Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00020476
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Sepsis
Keywords: presumed sepsis
MeSH Terms: conditions — Sepsis | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Open label -- 6 interval doses
  Interventions: Drug: piperacillin-tazobactam

INTERVENTIONS:
Drug: piperacillin-tazobactam — 6 doses intravenously at the following doses:
  Infants <32 weeks gestation at birth < 14 days PNA 100 mg/kg Q8 ≥ 14 weeks PNA 100 mg/kg Q6
  Infants ≥32 weeks gestation at birth < 14 days PNA 100 mg/kg Q6
  ≥ 14 days PNA 100 mg/kg Q6

SUMMARY:
This is a phase I open label multi-dose study to investigate the pharmacokinetics and safety of piperacillin-tazobactam in infants < 61 days of age with suspected sepsis. There will be four cohorts of 8 infants each:

1. < 32 weeks gestational age (GA) and < 14 days postnatal age (PNA)
2. < 32 weeks gestational age and >=14 days postnatal age
3. >=32 weeks gestational age and < 14 days postnatal age
4. >=32 weeks gestational age and >=14 days postnatal age. The study requires administration of 6 doses of study drug along with other antimicrobials per standard of care followed by 1 week of safety monitoring. Four 200 µL pK samples will be obtained at steady state. The risks are reasonable vs. the benefits and have been minimized appropriately. There may be benefit to the subjects (administration of broad spectrum empirical antimicrobial therapy), and information from the study may benefit a large number of other infants in whom the drug is currently being administered despite the lack of PK data in this population.

DETAILED DESCRIPTION:
Procedures Prior to Receipt of First Dose of Study Drug

Parental/Guardian Permission Prior to the start of any study-related procedure, a signed and dated informed consent and HIPAA authorization must be obtained and documented in the infant's medical record. Once it has been determined that the infant meets all inclusion criteria and no exclusion criteria, the infant will be assigned a subject identification number that will be used on the subject's CRFs and will be considered enrolled.

Study Drug Administration

Assignment to Therapy Groups Infants meeting the eligibility will receive piperacillin-tazobactam. Concomitant use of an aminoglycoside is suggested. Enrollment and study drug dose will be stratified by GA and PNA. After enrollment information for the eligible infant is provided, the dosage assignment and subject number will be allocated. If an infant is assigned a study drug and a number, but does not receive study drug, the subject number will not be used again. The reason for not dosing the subject will be noted on the case report form (CRF).

Dosing:

Infants <32 weeks gestation at birth

< 14 days PNA 100 mg/kg Q8

>=14 weeks PNA 100 mg/kg Q6

Infants ≥32 weeks gestation at birth

< 14 days PNA 100 mg/kg Q6

>=14 days PNA 100 mg/kg Q6

Dispensing of Study Drug The pharmacist at each site will prepare and dispense the study drug. Study drug will be dispensed by the pharmacy in appropriate size syringes and administered via a syringe pump at a rate calculated based on the infants' body weight in kilograms (kg) per local standard of care, but with a target of infusing the product over 30 minutes. Immediately following study drug administration the infusion tubing will be flushed per the unit protocol.

Piperacillin-tazobactam should not be mixed with or physically added to solutions containing other drugs. Infusion vials of piperacillin-tazobactam will be reconstituted and stored per the package insert and local pharmacy requirements. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration, whenever solution and container permit.

Dosing for infants receiving piperacillin-tazobactam per local standard of care Once an infant is enrolled in the study, steady state PK levels may be drawn after the 4th, 5th, or 6th dose of piperacillin-tazobactam. These doses may include both pre-study doses of piperacillin-tazobactam and post-consent, 'on-study', doses if the dosage and dosing interval of piperacillin-tazobactam remains the same. If a subject receives < 4 doses of on-study piperacillin-tazobactam at the time of steady state PK sampling, ≥ 4 doses (pre-study doses + on study doses) of piperacillin-tazobactam should be recorded on the Study Drug Administration CRF.

Other antimicrobial treatments Investigators are encouraged to provide infants with concomitant aminoglycoside therapy. Use of other antimicrobial agents (vancomycin, antifungals) may be given per local standard of care. A maximum of 6 doses of on study piperacillin-tazobactam will be administered under this protocol. Additional doses piperacillin-tazobactam or other antimicrobials may be administered per standard of care but will not be recorded on study CRFs.

Procedures by Visit

Pre-Study Drug Administration Procedures (Study Day 0)

The following procedures will be completed prior to the administration of study drug:

a. Review of Inclusion/Exclusion Criteria prior to infant enrollment b. Obtain signed and dated informed consent/HIPAA consent. c. Collect demographic data and medical history d. Perform a complete physical examination e. Obtain and record infant weight and medication dosing weight for calculation of appropriate study drug dose if different from actual weight f. Record results from hematology and serum chemistry labs if obtained within 72 hours prior to enrollment in accordance with local standard of care. Use the laboratory values closest to enrollment if there have been multiple tests.

1. Hematology labs will include: hematocrit, hemoglobin, white blood cell count with differential, and platelet count.
2. Serum chemistry will include glucose, creatinine, blood urea nitrogen, aspartate transaminases (AST), alanine transaminase (ALT), alkaline phosphatase, total and direct bilirubin, sodium, potassium, chloride, calcium, magnesium, total protein, and albumin.

g. Record results of sterile body fluid cultures (blood, urine, CSF, peritoneal fluid) obtained as standard clinical care in the 72 hours prior to study drug administration. Record urine cultures only if obtained by sterile catheterization or suprapubic aspiration.

h. Document concomitant medications in the 72 hours prior to study drug administration.

Procedures During Study Drug Administration (Study Days 1-2)

a. Record study drug timing of infusion before the PK samples are obtained - this includes start/stop times of infusion and amount given b. Assess and record AEs from the time of the first dose of study drug. c. Assess and record SAEs from the time of the first dose of study drug. d. Record all concomitant antimicrobials and vasopressors administered e. Collect blood for PK analysis (Appendix 2) f. Record result for clinical laboratory assessments obtained per local standard of care one time daily while on study drug.

1. Hematology assays will include: hematocrit, hemoglobin, white blood cell count with differential, and platelet count.
2. Serum chemistry will include glucose, creatinine, blood urea nitrogen, aspartate transaminases (AST), alanine transaminase (ALT), alkaline phosphatase, total and direct bilirubin, sodium, potassium, chloride, calcium, magnesium, total protein, and albumin.

g. Record the results of cultures from sterile body fluids (blood, urine, CSF, peritoneal fluid, or any other sterile body fluid) as obtained per standard of care. Record urine cultures only if obtained by sterile catheterization or suprapubic aspiration.

Procedures following Study Drug Administration

1. Assess and record adverse events (AEs) for 72 hours following the last dose of study drug
2. Assess and record serious adverse events (SAEs) for 7 days following the last dose of study drug

Safety

Adverse Events

Reporting period AEs will be recorded from the time of informed consent until 72 hours following the last dose of study drug for non SAEs and until 7 days after the last dose of study drug for SAEs. Any AE that occurs between the time informed consent is obtained and the initial dose of study, that is considered related to a protocol specified procedure, must be reported.

Procedures for assessing, recording and reporting AEs Throughout the duration of the study, the investigator will closely monitor each subject for clinical evidence of drug intolerance and monitor all clinically obtained laboratory values for laboratory evidence of AEs. AEs not explained by the infant's underlying illness which occur during the course of the study will be reported in detail on the appropriate CRFs and followed until resolution or until it becomes stable. All SAEs will be reported to study's medical monitor within 24 hours.

The description of the AE will include description of event, start date, stop date, intensity, if it was serious, and relationship to the study drug. The investigator must verify this information.

The Investigator is responsible for assessing relationship to study medication.

Blood Volume for PK and Safety Laboratory Tests

Blood sample volume will be minimized by:

Hematology and chemistry laboratory measures will be recorded from laboratories drawn as standard of care and will not be drawn strictly for purpose of this study.

A limited PK sampling scheme will be employed such that no more than a total of 0.8 mL of blood (4 samples) is obtained from each subject for PK analysis.

Statistical Methods

Definitions and Populations for Analysis All infants who receive piperacillin-tazobactam will be analyzed. These infants will comprise the population for the safety analysis, and if any PK samples are obtained, their blood will be evaluated in the PK analysis.

Demographics Descriptive statistics such as number of observations, mean, median, 95% confidence interval, standard deviation, standard error, minimum, and maximum will be presented by group for continuous variables (such as age, weight, etc). Other descriptive statistics such as counts, proportions, and/or percentages will be presented by dosage group to summarize discrete variables (such as race, sex, success rates, mortality rates, etc.) The number of infants completed, and discontinued early from study, and the reasons for discontinuation, will be summarized. Demographic and baseline characteristics will be summarized by group. Variables include race, age, sex, and selected clinical variables recorded prior to initiation of study drug.

7.4 Pharmacokinetics

The following PK parameters will be estimated:

1. Systemic clearance (CL)
2. Volume of distribution (Vd)
3. maximum concentration (Cmax), time at maximum concentration (Tmax), area under the curve (AUC0-Τ), Ke and half-life (t1/2)
4. CSF/plasma piperacillin-tazobactam concentration ratio
5. Endotracheal aspirate/plasma piperacillin-tazobactam concentration ratio
6. Saliva/plasma piperacillin-tazobactam concentration ratio
7. Urine/plasma piperacillin-tazobactam concentration ratio

The PK parameters and MIC will be used to estimate pharmacodynamic parameters of exposure (time above MIC). Using sparse sampling PK analysis, parameters (clearance, Vd) will be estimated for the following each of the cohorts. The plasma concentrations-time profiles of piperacillin-tazobactam will be presented in tabular and graphical form by subject, age cohort, and dosage level. The relationship between plasma concentrations and/or PK parameters with demographic factors (weight, gestational age, postnatal age), disease severity, toxicity and co-administered medications will be investigated. Analysis of potential relationships between drug and exposure in subjects and the resulting efficacy and/or safety response will be conducted.

Sample Size The sample size is designed to assess multiple dose PK of piperacillin-tazobactam in young infants. At least 4 infants will be enrolled in each of the GA/PNA cohorts. Infants will be enrolled to ensure that at least 4 infants with ≥3 evaluable PK samples are enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Written permission from parent or legal guardian
2. < 61 days of age
3. Likely to survive beyond the first 48 hours after enrollment
4. Sufficient intravascular access (either peripheral or central) to receive study drug.

AND ONE OF THE FOLLOWING

1. Suspected systemic infection
2. Receiving piperacillin-tazobactam as part of standard of care

Exclusion Criteria:

1. History of allergic reactions to any penicillin, cephalosporins, or beta-lactamase inhibitors
2. Urine output < 0.5 mL/hr/kg over the prior 24 hours
3. Serum creatinine > 1.2 mg/dL
4. Any condition which would make the subject or the caregiver, in the opinion of the investigator, unsuitable for the study

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip B. Smith, MD, Principal Investigator — Duke Universtity Medical Center
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - Children's Mercy Hospital, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Cohen-Wolkowiez M, Benjamin DK Jr, Ross A, James LP, Sullivan JE, Walsh MC, Zadell A, Newman N, White NR, Kashuba AD, Ouellet D. Population pharmacokinetics of piperacillin using scavenged samples from preterm infants. Ther Drug Monit. 2012 Jun;34(3):312-9. doi: 10.1097/FTD.0b013e3182587665. PMID 22569355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants recruited from intensive care nurseries.First subject was recruited/enrolled on 1/29/2010. Last subject was enrolled on 7/29/2010. A total of 32 subjects were enrolled at 4 participant sites.
Groups:
- GA of 32 Wks, PNA of 14 Days: Open label -- 6 interval doses
  piperacillin-tazobactam : 6 doses intravenously at the following doses:
  Infants <32 weeks gestation at birth < 14 days postnatal age (PNA) 100 mg/kg Q8 ≥ 14 weeks PNA 100 mg/kg Q6
  Infants ≥32 weeks gestation (GA) at birth < 14 days PNA 100 mg/kg Q6
  ≥ 14 days PNA 100 mg/kg Q6
Period: Overall Study
Arm/Group | GA of 32 Wks, PNA of 14 Days
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GA of 32 Wks, PNA of 14 Days: Open label -- 6 interval doses
  piperacillin-tazobactam : 6 doses intravenously at the following doses:
  Infants <32 weeks gestation at birth < 14 days PNA 100 mg/kg Q8 ≥ 14 weeks PNA 100 mg/kg Q6
  Infants ≥32 weeks gestation at birth < 14 days PNA 100 mg/kg Q6
  ≥ 14 days PNA 100 mg/kg Q6
Arm/Group | GA of 32 Wks, PNA of 14 Days
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.1 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Piperacillin Pharmacokinetics (PK)
Description: To study how Piperacillin is metabolized in the body by measuring the drug concentration in plasma samples collected at different time points during the study
Time Frame: 2-3 days after infant receives 1st drug dosing
Population: All 32 subjects that were enrolled during the study.
Measure: Median (95% Confidence Interval); unit: L/hr/kg
Groups:
- PK Analysis Cohort - Piperacillin Plasma Clearance: Open label -- 6 interval doses
  piperacillin-tazobactam : 6 doses intravenously at the following doses:
  Infants <32 weeks gestation at birth < 14 days PNA 100 mg/kg Q8 ≥ 14 weeks PNA 100 mg/kg Q6
  Infants ≥32 weeks gestation at birth < 14 days PNA 100 mg/kg Q6
  ≥ 14 days PNA 100 mg/kg Q6
Arm/Group | PK Analysis Cohort - Piperacillin Plasma Clearance
Number analyzed (Participants) | 32
L/hr/kg | 0.0799 [0.0677 to 0.093]

ADVERSE EVENTS:
Description: AEs/SAEs were collected. None SAE was observed.
Arm/Group | GA of 32 Wks, PNA of 14 Days
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes